CLINICAL TRIAL: NCT06697067
Title: The Comparison of Interrupted Modified Smead-Jones Versus Conventional Continuous Suturing Technique for Closure of Rectus Sheath in Patients Undergoing Laparotomy for Hollow Viscus Perforation.
Acronym: Farrukh 24
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Edward Medical University (Other)
Collaborators: Mayo Hospital Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 163/RC/Kemu; 12921/REG/KEMU/24 (Other: ASRB, King Edward Medical University, Lahore.)
Record Dates: First submitted 2024-11-17; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Wound Dehiscence, Surgical
Keywords: Farrukh 24
MeSH Terms: conditions — Surgical Wound Dehiscence

STUDY DESIGN:
Intervention Model Description: Randomised control trials
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient undergoing emergent laparotomy due to hollow viscus perforation (Experimental)
  Interventions: Procedure: modified smead jones
- patient undergoing emergent laparotomy (Experimental): patient undergoing emergent laparotomy for hollow viscus perforation
  Interventions: Procedure: conventional comtinuous suture techniques

INTERVENTIONS:
Procedure: modified smead jones — interrupted suture technique
  Arms: Patient undergoing emergent laparotomy due to hollow viscus perforation
Procedure: conventional comtinuous suture techniques — continuous suture technique
  Arms: patient undergoing emergent laparotomy

SUMMARY:
After taking approval from Board of Studies, IRB & ASRB of KEMU, 108 patients fulfilling inclusion criteria will be admitted in Department of General Surgery, East Surgical Ward, Mayo Hospital Lahore through Emergency Department. Firstly patients will be seen in emergency department, history and clinical examination will be done and laboratory investigations and imaging will be done. All the patients aged greater than 18 years undergoing emergency laparotomy for hollow viscus perforation will be included in the study. Informed consent will be obtained. Demographic data including name, age, sex will be recorded.

Emergency laparotomy will be done with midline incision and intra-operative findings will be recorded. Thorough peritoneal lavage will be done and necessary procedures will be carried out for the pathology identified, and abdominal drains will be placed. The patients then will be randomly divided into 2 groups; group A (Experimental Group) undergoing Modified Smead-Jones interrupted suture technique and group B (Reference Group) undergoing conventional continuous suture closure of rectus sheath. In Modified Smead-jones suture technique describe as a far bite starting at 2 cm on the edge of linea from outside-in and then taking a near bite of 0.5 cm on the other side inside-out- a near bite on the same side outside-in and then a far bite on the other side inside-out. The suture was next converted to a horizontal mattress by taking a far bite 1 cm above or below the previous bite on the other side- near bite on the same side, near bite on the other side, and finally a far bite on the same side. The two ends of the suture were tied to approximate the edges of the linea alba9. In conventional continuous closure suture technique I will use number 1 polypropylene suture, care being taken to place each bite 1-1.5 cm from the cut edge of linea alba and successive bites being taken 1cm away from each other The edges of linea alba were gently approximated without strangulation with an attempt to keep a suture to wound length ratio of 4:110.Rectus sheath will be closed by the suture material No.1 polypropylene in both groups.

The midline laparotomy wound will be managed with daily antiseptic dressing and intravenous antibiotics. All patients will be examined daily till discharge then weekly till 2 weeks and on each visit, a slandered physical examination of abdomen of wound will be done and presence of burst abdomen will be noted. When there are no signs of burst abdomen (after 14 postoperative days) the laparotomy wound will be considered normal. All the data will be collected in accordance to patient's proforma.

DETAILED DESCRIPTION:
An emergency laparotomy is a common surgical procedure, performed for a wide variety of intra-abdominal pathologies, which has a significant associated morbidity and mortality. Each year, approximately 30,000 emergency laparotomies are performed in the UK [1]. A major surgical complication after emergency midline laparotomy is abdominal fascial dehiscence. Dehiscence is associated with increased morbidity and mortality rates up to 30%, prolonged hospital stay, and a long-term risk of developing incisional hernia [1].

Hollow viscus perforation is one of the most common cause of peritonitis necessitating emergency surgical intervention. The diagnosis is mainly based on clinical grounds. Plain abdominal X-rays (erect) may reveal dilated and edematous intestines with pneumoperitoneum. Local findings include abdominal tenderness, guarding or rigidity, distension, diminished bowel sounds and systemic findings include fever, chills or rigor, tachycardia, sweating, tachypnea, restlessness, dehydration, oliguria, disorientation and ultimately shock. Exposure of the normally sterile peritoneal cavity to intraluminal contents causes secondary bacterial peritonitis. The peritoneal contamination due to bowel perforation is one of the leading risk factor for occurrence of burst abdomen [2].

Laparotomy wound dehiscence (LWD) is a term used to describe separation of the layers of a laparotomy wound before complete healing has taken place. Other terms used interchangeably are acute laparotomy wound failure and burst abdomen. Frequency of laparotomy wound dehiscence in the relevant literature is cited in the range of 0.2% to 10%[3,4]. The occurrence of fascial dehiscence represents a risk factor for increased mortality rates of up to 25%[5] [11] [12] Acute wound failure may be occult or overt, partial or complete. Overt wound failure follows early removal of sutures leading to evisceration. Occult dehiscence occurs with disruption of musculo-aponeurotic layer beneath intact skin sutures. Wound dehiscence has been noted to occur when a wound fails to gain sufficient strength to withstand stresses placed upon it. The separation may occur when overwhelming forces break sutures, when absorbable sutures dissolve too quickly or when tight sutures cut through tissues [6].

Conventional continuous closure technique has been shown to compromise blood supply and thereby poor wound holding, during initial phases of wound dehiscence. Surgeons have been continuously striving to overcome postoperative complications associated with laparotomy wound closure using newer techniques and newer suture materials. Several reviews have studied the optimal suture repair for closing the abdominal fascia, but no consensus has been reached. Hence, it is imperative for us to ascertain better method of closing the abdomen. While the choice may not be so important in elective patients who are nutritionally adequate, do not have any risk factor for dehiscence and are well prepared for surgery, however it may prove crucial in emergency patients who often have multiple risk factors for developing dehiscence and the strangulation of the sheath is the proverbial last straw in precipitating wound failure Majority of the studies suggest that, the most effective method of midline abdominal fascial closure in the elective setting is mass closure incorporating all layers of abdominal wall except skin in continuous technique with No. 1 or 2 delayed absorbable monofilament suture material with suture length to wound length ratio 4:14-7 .Many randomized controlled trials showed that odds of the burst abdomen are reduced with the interrupted method of closure as compared to continuous.

A study done by AGHARA CB et al8 to compare incidence of burst abdomen between modified smead-jones interrupted suture technique (2%) versus conventional continuous closure (14%) in patient undergoing hollow visus perforation. However the previous done studies have not taken into account a specific population with specific risk factor to compare these two suturing techniques so the aim of present study is to compare the incidence of burst abdomen in the patient undergoing midline abdominal wall closure with modified smead jones interrupted suture9 techniques (Experimental group) and conventional continuous suturing technique10 (Reference Group) in patient undergoing emergency laparotomy for hollow viscus perforation.

ELIGIBILITY:
Inclusion Criteria:All patients of both genders with age greater than 18 to 60 years, undergoing emergency laparotomy through midline incision for hollow viscus perforation.

ASA grade III -

Exclusion Criteria:Patients who had undergone a previous laparotomy for any condition or had an incisional hernia or burst abdomen at presentation.

Patients undergoing laparotomy with anterior abdominal wall injury in the form of muscle, hematoma, disruption or abdominal wall laceration.

-

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Estimated)
Dates: Start 2024-06-06 (Actual); Primary Completion 2025-06-06 (Estimated); Study Completion 2025-06-21 (Estimated)

PRIMARY OUTCOMES:
safety | 15days after emergent laparotomy
  best closure technique of rectus sheath

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, King Edward Medical University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
still under consideration